CLINICAL TRIAL: NCT00004024
Title: Immunotherapy for Malignant Glioma - Phase II Trial of Autologous Cancer Antigen Specific Immunotherapy
Brief Title: Biological Therapy Following Surgery and Radiation Therapy in Treating Patients With Primary or Recurrent Astrocytoma or Oligodendroglioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067243; P30CA022453 (NIH); WSU-C-1403-BT; NCI-G99-1567; NCT00004018 (obsolete NCT alias); NCT00004019 (obsolete NCT alias); NCT00004020 (obsolete NCT alias); NCT00004021 (obsolete NCT alias); NCT00004023 (obsolete NCT alias)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult subependymoma; adult oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma; adult diffuse astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma, Subependymal; Gliosarcoma | interventions — aldesleukin; FANG vaccine; Muromonab-CD3; sargramostim; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: aldesleukin
Biological: autologous tumor cell vaccine
Biological: muromonab-CD3
Biological: sargramostim
Biological: therapeutic autologous lymphocytes
Procedure: surgical procedure
Radiation: radiation therapy

SUMMARY:
RATIONALE: Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing. Combining different types of biological therapies may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of biological therapy following surgery and radiation therapy in treating patients who have primary or recurrent astrocytoma or oligodendroglioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of immunotherapy with irradiated autologous tumor cell vaccine and adoptive immunotherapy, in terms of time to progression and median and one-year survival, in patients with primary or recurrent malignant astrocytoma or oligodendroglioma.
* Determine the immunogenicity of malignant gliomas in patients treated with this regimen.

OUTLINE: Patients are stratified according to extent of disease, extent of antigen-specific response to vaccination, performance status (0 vs 1), prior therapy (yes vs no), and gender.

Patients undergo tumor resection on week 1. Patients without recurrent disease receive local radiotherapy on weeks 2-8. Beginning week 10-12, patients are vaccinated with irradiated autologous tumor cells and sargramostim (GM-CSF) and then receive GM-CSF alone intradermally at vaccination sites daily for 4 days. Patients are revaccinated 4 weeks later and may receive up to 3 additional vaccinations every 2 weeks until a response is detected.

Patients undergo peripheral blood mononuclear cell collection on week 14 followed by monoclonal antibody OKT3-activated T lymphocytes IV over 1-6 hours with alternating interleukin-2 IV once every other day for 5 doses over 10 days beginning on week 16. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients may receive one additional course of immunotherapy as above.

Patients are followed at 1 week, monthly for 3 months, every 3 months for 2 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven grade II, III, or IV astrocytoma or oligodendroglioma

  * Evidence of primary or recurrent tumor by MRI
  * Resectable disease

    * At least 20,000,000 viable cells obtained from surgical specimen for use in the immunization part of this study

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* SWOG 0 or 1

Life expectancy:

* At least 6 months

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least lower limit of normal
* No active or recent uncontrolled bleeding

Hepatic:

* Bilirubin normal
* SGOT no greater than 2 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)

Renal:

* Creatinine normal

Other:

* Able to be weaned off steroids
* Negative stool guaiac
* No impaired immunity
* No uncontrolled diabetes
* No active uncontrolled infections
* No other serious disease
* No other malignancies within the past 5 years except curatively treated basal or squamous cell skin cancer or carcinoma in situ of the cervix
* No psychological, familial, sociological, or geographical conditions that would preclude compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No concurrent chemotherapy except for progressive disease

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* Radium implants allowed

Surgery:

* Not specified

Other

* At least 1 week since prior therapy and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 1997-06; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew E. Sloan, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- [Result] Sloan AE, Dansey R, Zamorano L, Barger G, Hamm C, Diaz F, Baynes R, Wood G. Adoptive immunotherapy in patients with recurrent malignant glioma: preliminary results of using autologous whole-tumor vaccine plus granulocyte-macrophage colony-stimulating factor and adoptive transfer of anti-CD3-activated lymphocytes. Neurosurg Focus. 2000 Dec 15;9(6):e9. doi: 10.3171/foc.2000.9.6.10. PMID 16817692